CLINICAL TRIAL: NCT05510986
Title: The Effect of Oxycodone Hydrochloride on Catheter-related Bladder Discomfort After TURBT Under General Anesthesia
Brief Title: The Effect of Oxycodone Hydrochloride on CRBD After TURBT Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: lingzi-2022-1
Record Dates: First submitted 2022-08-02; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Effect of Drug; Adverse Effect of Opioids
Keywords: Oxycodone Hydrochloride; CRBD; TURBT; general anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl group (Active Comparator): Drugs
  Interventions: Drug: Fentanyl group
- Oxycodone Hydrochloride group (Experimental): Drugs
  Interventions: Drug: Oxycodone Hydrochloride group

INTERVENTIONS:
Drug: Fentanyl group — Dilute fentanyl hydrochloride injection (1ml:0.1mg) with 0.9% normal saline to 10μg/ml, 1μg/kg fentanyl is slowly injected intravenously 10 minutes before the end of the operation, and the administration speed is not less than 5 minutes.
  Other Names: Active Comparator
  Arms: Fentanyl group
Drug: Oxycodone Hydrochloride group — Dilute Oxycodone Hydrochloride injection (1ml:10mg) with 0.9% normal saline to
  1mg/ml, 0.1mg/kg Oxycodone Hydrochloride is slowly injected intravenously 10 minutes before the end of the operation, and the administration speed is not less than 5 minutes.
  Other Names: Experimental
  Arms: Oxycodone Hydrochloride group

SUMMARY:
The purpose of this study is to investigate the effect of Oxycodone Hydrochloride on catheter-related bladder discomfort in patients undergoing transurethral resection of bladder tumor after general anesthesia.

DETAILED DESCRIPTION:
Catheter-related bladder discomfort(CRBD) is a frequent complication after indwelling catheter under general anesthesia. The incidence of CRBD in patients undergoing Transurethral resection is as high as 66.7-91.2%.CRBD may lead some poor prognosis including postoperative restlessness, bleeding, and circulatory instability.therefore，how to reduce the incidence of CRBD is one of the urgent problems to be solved in clinic.

Oxycodone Hydrochloride is a strong opioid receptor agonist used in clinic at present. It has certain advantages in the regulation of visceral pain and can produce analgesic effect without causing restlessness, gastrointestinal motility inhibition and respiratory inhibition through stimulating the μ and κ opioid receptor simultaneously. However, the effect of Oxycodone Hydrochloride on catheter-related bladder discomfort in patients undergoing transurethral resection of bladder tumor after general anesthesia is still unknown. The purpose of this study is to explore whether Oxycodone Hydrochloride via intravenous injection could reduce the incidence of CRBD in patients undergoing transurethral resection of bladder tumor after general anesthesia and could not increase other complications during the recovery period of general anesthesiathe.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old;
* ASA I - III;
* Plan to perform transurethral resection of bladder tumor under general anesthesia; (
* Agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Refuse to participate in this study;
* Emergency surgery;
* Catheter was indwelling before operation;
* Taking opioids for a long time before operation;
* Previous history of schizophrenia, epilepsy, Parkinson's disease or myasthenia gravis;
* Unable to communicate due to coma, severe dementia or language disorder before operation;
* Critical condition (ASA grade ≥ IV before operation); Severe renal function damage (requiring renal replacement therapy); Severe liver function damage (child Pugh grade C); Acute stage of chronic obstructive pulmonary disease, severe asthma, severe pulmonary heart disease;
* History of opioid allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of catheter-related bladder discomfort | 1 hour
  CRBD is symptoms vary among patients from burning sensation and pain in the suprapubic and penile areas to urinary urgency.
  4 grades 0:No discomfort
  1. Mild discomfort only reported upon questioning
  2. Moderate discomfort, urge to pass urine reported by the patient without questioning
  3. Severe discomfort, urge to pass urine accompanied by behavioral responses, such as flailing limbs, strong verbal responses, or attempt to pull out the catheter

SECONDARY OUTCOMES:
The incidence of Nausea and vomiting | 1 hour
  Nausea refers to patients who have gastrointestinal symptoms but do not spit out stomach contents. Vomiting means that the patient has gastrointestinal symptoms and vomits stomach contents
Degree of sedation | 1 hour
  Ramsay evaluation
Degree of pain | 1 hour
  NRS
the incidence of other complication | 1 hour
  Respiratory depression, itching, shivering

CONTACTS AND LOCATIONS:
Overall Officials: Ni xinli, MD, Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No